CLINICAL TRIAL: NCT06922578
Title: Clinical and Radiographic Success of Pulpotomy Using Neoputty Mineral Trioxide Aggregate Versus Pulpectomy Using Endoflas In Primary Molars With Irreversible Pulpitis: A Randomized Controlled Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Manar Motawie Abdulfattah, DR., Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Neoputty MTA pulpotomy
Record Dates: First submitted 2025-04-03; First posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Pulpitis - Irreversible

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neoputty MTA pulpotomy (Experimental)
  Interventions: Procedure: NeoPUTTY MTA pulpotomy
- Endoflas pulpectomy (Experimental)
  Interventions: Procedure: Endoflas pulpectomy

INTERVENTIONS:
Procedure: NeoPUTTY MTA pulpotomy — Neoputty MTA pulpotomy performed in vital primary molars with symptomatic irreversible pulpitis
  Arms: Neoputty MTA pulpotomy
Procedure: Endoflas pulpectomy — Endoflas pulpectomy in vital primary molars with symptomatic irreversible pulpitis
  Arms: Endoflas pulpectomy

SUMMARY:
The goal of this randomized clinical trial is to evaluate the clinical and radiographic success of pulpotomy using Neoputty MTA vital primary molars diagnosed with symptomatic irreversible pulpitis.

The main question it aims to answer is:

Will Neoputty MTA pulpotomy have higher clinical and radiographic success in comparison to Endoflas pulpectomy in primary molars with irreversible pulpitis?

ELIGIBILITY:
Inclusion Criteria:

* Children with spontaneous pain lasting a few seconds to several hours.
* Pain is intensified by thermal stimulus and persists after its removal.
* Pulp hemorrhage after performing access cavity and deroofing of pulp chamber showing reddish pink healthy pulp tissue.
* Radicular pulp health is verified by achieving hemostasis within six minutes of compression using a cotton pellet with 2% sodium hypochlorite.
* Absence of peri-apical or inter-radicular radiolucency, widening of periodontal ligament space, internal or external root resorption.

Exclusion Criteria:

* Unrestorable primary molars.
* Primary molars with uncontrolled pulp hemorrhage or pulp necrosis.
* Medically compromised patients who have systemic disease.
* Uncooperative children who refuse treatment.

Ages: 4 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 66 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
postoperative pain | within 24 hours, after 1 week, 3, 6, 9, and 12 months
  postoperative pain will be assessed using the visual analogue scale (VAS) within 24 hours, after 1 week, 3, 6, 9, and 12 months. The patients are asked to point to the face that best represents how they are feeling at the follow-up visits.

CONTACTS AND LOCATIONS:
Overall Officials: DR, Principal Investigator — assistant lecturer

IPD SHARING:
Plan to Share IPD: No